CLINICAL TRIAL: NCT04345484
Title: Action for Positive Brain Health Now: Ready, Set, Go
Brief Title: Action for Brain Health Now: Ready, Set, Go
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Nancy Mayo, Nancy Mayo, Principal Investigator, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-6202
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Hiv
Keywords: Cognition; Exercise; Goal-setting; Intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMT Intervention + Health Lifestyle Program (Experimental): The intervention group will participate in GMT, a standardized cognitive rehabilitation program which will be given as per the manual and which consists of 9 sessions each 2-hours in duration. They will also participate in the Healthy Lifestyle Program (HLP), which includes physical activity monitoring (step count, calories burned and sleep) with the Garmin vívofit 4 Activity Tracker, and recording and monitoring of goals with the My Goals app. Moreover, participants will be offered an exercise program with weaning to community-based resources and home exercise recommendations for longer-term sustainability.
  Interventions: Behavioral: Goal-management training
- Health Lifestyle Program (Active Comparator): The control group enters directly into the HLP without any other study visits. The HLP includes physical activity monitoring (step count, calories burned and sleep) with the Garmin vívofit 4 Activity Tracker, and recording and monitoring of goals with the My Goals app. Moreover, participants will be offered an exercise program with weaning to community-based resources and home exercise recommendations for longer-term sustainability.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Goal-management training — 9-week goal-management program
  Arms: GMT Intervention + Health Lifestyle Program
Behavioral: Control — Healthy Lifestyle Program
  Arms: Health Lifestyle Program

SUMMARY:
HIV (human immunodeficiency virus) can have subtle but important effects on the brain, leading to difficulties in memory, concentration, or problem solving. Goal-setting interventions have been shown to help individuals maintain their physical activity in order to improve brain health. The study objective is to estimate the extent to which goal management training before a personalized healthy lifestyle program is associated with greater adherence to health recommendations, achievement of health-related goals, and better brain health and general health outcomes compared to the healthy lifestyle program alone. Participants will be randomized to either Goal Management Training (GMT) and a Healthy Lifestyle Program (HLP) or the control group (HLP alone).

DETAILED DESCRIPTION:
Based on healthy aging research in HIV- populations, it is already known that many older people living with HIV could protect or improve their brain health through lifestyle change . However, no intervention is effective if it is not done. Sustained lifestyle change is hard for everyone, but expected to be harder still for those with a chronic condition that affects cognitive ability, eroding the very executive functions needed for effective goal-directed behavior. Thus, the key question is not whether interventions will help brain health in HIV but rather how we can improve adherence to the most promising interventions in people experiencing brain health challenges.

This study will test an innovative approach to enhance adherence to lifestyle interventions, building on feasibility evidence from pilot trials in the Brain Health Now (BHN) study. Goal Management Training (GMT) is a fully manualized cognitive rehabilitation program delivered over 9 weeks in small groups. It targets executive dysfunction, teaching self-management and mindfulness. GMT also trains participants to use explicit strategies to reduce cognitive load in everyday tasks, and methods to cue attention to maintain focus on specific tasks, through weekly 2-h sessions and practice at home. We hypothesize that GMT priming before a personalized Healthy Lifestyle Program (HLP) will improve adherence to that program and subsequently improve health outcomes, compared to the HLP without GMT priming, in cognitively frail men and women living with HIV.

Study objectives

The overall objective of Action for Brain Health Now is to understand, empower and act to protect and improve brain health in HIV, in order to empower patients to take charge of their brain health. This sub-study is directed to the third aim, act. This proposed study addresses the real-world challenge of implementing tailored recommendations, recognizing that the cognitively frail individuals who would benefit the most from lifestyle changes are least equipped to successfully adopt and sustain healthy behaviours. We will trial a novel cognitive rehabilitation approach using goal-management training to boost adherence to a tailored active living intervention.

Specific objective

Estimate the extent to which cognitive rehabilitation before a personalized healthy lifestyle program (HLP) is associated with greater uptake of health recommendations, achievement of health-related goals, and better brain health and general health outcomes compared to the HLP alone.

Methods

Design

A blinded, randomized control trial will be conducted in 100 participants at two sites (Montreal and Vancouver) in order to assess the impact of cognitive rehabilitation on the uptake of a healthy lifestyle program. More specifically, 50 participants will be recruited in Montreal and 50% (i.e. 25 participants) will be assigned to the intervention group and the other 50% (i.e. 25 participants) will be assigned to the control group. The same is true for the site in Vancouver.

Recruitment

The eligibility criteria will be given to the data team who will do a search among the participants and send the investigators a list of ID of potential participants. If these potential participants have agreed, in the main study consent form, to be contacted for sub-studies, they will get a phone call, email or will be contacted directly during a clinic visit by the research coordinator involved in the main study (ABHN). Ethics approval for the Glen site including Royal Victoria Hospital & Center for Innovative Medicine (CIM) / Montreal, the Clinique Médicale l'Actuel / Montreal and Clinique Médicale Urbaine Quartier Latin / Montreal will be obtained through the MUHC REB. A separate application for the university-based clinic at St-Paul's Hospital / Vancouver will be sent to their own REB for approval.

Intervention

The sample will be drawn from cohort participants. The ABHN full cohort will receive a personalized My Personal Brain Health Dashboard populated directly from their study data accompanied by a document with 7 Simple Tips for Better Brain Health. In addition, the participants of this trial will receive a short list of relevant local resources (e.g. low-cost gyms, community social groups, smoking cessation programs). To test whether a cognitive rehabilitation program will increase healthy lifestyle adherence, people meeting eligibility criteria will be identified and, if in Vancouver or Montreal, offered entry into a randomized trial asking whether priming with GMT will increase adherence to a HLP focused on physical and social activity. All of the participants who agree to enter the trial will be invited to attend the Ready, Set Workshop which will occur before randomization at each site (50 participants per site) and will last approximately four hours long.

Ready: All of the participants will be shown how to best interpret the My Personal Brain Health Dashboard. All of the participants will also be provided with the Garmin vívofit 4 Activity Tracker (worn on the wrist); they will also be trained how to use the Garmin vívofit 4 Activity tracker as well as the mobile app that accompanies it, the SmartAge digital platform for activity tracking and feedback (collaborator Guaraldi). Participants who do not have an app compatible device will be provided with one for the duration of the study.

Set: During the Workshop there will be instruction on SMART goals and demonstration of the My Goals app to use for recording and monitoring goals.

Go: Following the workshop, the participants will be randomized to priming with GMT as they enter the HLP, or to entering the HLP directly. The study period will last 52 weeks for both groups. The intervention group will participate in GMT, a standardized cognitive rehabilitation program which will be given as per the manual, which consists of 9 sessions each 2-hours in duration. The control group enters directly into the HLP without any other study visits.

For all the participants, the HLP includes, physical activity monitoring (step count, calories burned and sleep) with the Garmin vívofit 4 Activity Tracker, and recording and monitoring of goals with the My Goals app. Moreover, participants will be offered an exercise program with weaning to community-based resources and home exercise recommendations for longer-term sustainability.

In addition, all participants will be assigned a HLP coach to facilitate the transition into using community resources to meet their goals. The HLP coach will provide feedback, encouragement, and suggestions for increasing activity via weekly phone or text interactions throughout the HLP via the SmartAge Digital Platform. The physical activity target will be current Canadian guidelines for older people (150 minutes per week of moderate to vigorous exercise, accumulated in bouts of at least 10 minutes), while the social activity target will be one social event per week. All the strategies in the HLP have evidence for effectiveness.

The participants will also be asked to track the progress of their goals on the MyGoals app and report their participation in any activities they do by taking a picture of something to represent the activity. A research assistant will record the details of the activity (when, what, if it was alone or in a group) and then the picture will be deleted.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ for at least 1 year
* Able to communicate adequately in either French or English
* Able to give written informed consent
* One or more indicators of cognitive frailty (B-CAM<20, C3Q <60%) OR those that do not meet the criteria of successful aging (<7 subscales of SF-36 ≥Canadian Norms)

Exclusion Criteria:

* Dementia (MSK-rating stage 3 or more-cognitive component only
* Life expectancy < 3 years or other personal factor limiting the ability to participate in follow-up
* Non-HIV-related neurological disorder likely to affect cognition
* Known active CNS opportunistic infection or hepatitis C requiring IFN treatment during the follow-up period
* Known psychotic disorder
* Current substance dependence or abuse within the past 12 months
* People who have a medical contraindication to moderate exercise (walking for 10 minutes)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity | 0 and 12 months
  Number of weeks in which physical activity guidelines are met (150 min of moderate to vigorous activity in bouts of 10 minutes)
Change in social activity | 0 and 12 months
  Number of weeks in which at least one organized social activity was attended

SECONDARY OUTCOMES:
Change in goal attainment | 0 and 12 months
  Measured by number and diversity of goals set and met
Change in physical Activity pattern | 0 and 12 months
  Measured by Garmin vívofit 4 Activity Tracker (daily step counts, time spent in various cadence bands, sitting time)
Change in general health perception | 0 and 12 months
  Measured using Visual Analogue Health States (minimum score: 0, maximum score: 10; higher scores indicate a better outcome)
Change in sleep | 0 and 12 months
  Measured using Visual Analogue Health States (minimum score: 0, maximum score: 10; higher scores indicate a better outcome)
Change in distress | 0 and 12 months
  Measured using Visual Analogue Health States (minimum score: 0, maximum score: 10; higher scores indicate a better outcome)
Change in pain | 0 and 12 months
  Measured using Visual Analogue Health States(minimum score: 0, maximum score: 10; higher scores indicate a better outcome)
Change in fatigue | 0 and 12 months
  Measured using Visual Analogue Health States(minimum score: 0, maximum score: 10; higher scores indicate a better outcome)
Change in depression | 0 and 12 months
  Measured using Visual Analogue Health States(minimum score: 0, maximum score: 10; higher scores indicate a better outcome)
Change in anxiety | 0 and 12 months
  Measured using Visual Analogue Health States(minimum score: 0, maximum score: 10; higher scores indicate a better outcome)
Change in quality of life | 0 and 12 months
  Measured using Visual Analogue Health States (minimum score: 0, maximum score: 10; higher scores indicate a better outcome)

OTHER OUTCOMES:
Change in energy/fatigue | 0 and 39 weeks
  Measured using the 36-Item Short Form Survey Instrument (SF-36) (minimum score: 0, maximum score: 100, where higher scores indicate a better outcome)
Change in mood | 0 and 39 weeks
  Measured using the 36-Item Short Form Survey Instrument (SF-36) (minimum score: 0, maximum score: 100, where higher scores indicate a better outcome)
Change in physical function | 0 and 39 weeks
  Measured using the 36-Item Short Form Survey Instrument (SF-36) (minimum score: 0, maximum score: 100, where higher scores indicate a better outcome)
Change in cognitive performance | 0 and 39 weeks
  Measured using Brief Cognitive Ability Measure (B-CAM) (minimum score: 0, maximum: 35 in English; minimum:0, maximum: 42 in French; higher scores indicate better cognitive performance)
Self-reported cognition | 0 and 39 weeks
  Measured using Communicating Cognitive Concerns questionnaire (C3Q) (minimum:0, maximum: 36, higher scores indicate better self-reported cognition)
Change in health-related quality of life | 0 and 39 weeks
  Measured using the EuroQol-5D (EQ-5D) which includes a health index score (minimum: 0, maximum: 1; higher scores indicate a better outcome) and a visual analog score (minimum:0, maximum: 100; higher scores indicate a better outcome)
Change in global quality of life | 0 and 39 weeks
  Measured using the Patient Generated Index (PGI) (minimum: 1, maximum: 10; higher scores indicate a better outcome)
Change in Cardiovascular Risk Score | 0 and 39 weeks
  Measured using the Framingham Cardiovascular Disease Risk Score (minimum: 0, maximum: 30; higher score indicates higher cardiovascular disease risk)
Change in social network size and quality | 0 and 39 weeks
  Measured using the Collaborative Research on Ageing in Europe Social Network Index (minimum: 0, maximum: 100; higher score indicates a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mayo, PhD, Principal Investigator — McGill University; Marie-Josée Brouillette, MD, Principal Investigator — McGill University; Lesley Fellows, PhD/MD, Principal Investigator — McGill University
Locations (4):
- Canada (4):
  - The John Ruedy Immunodeficiency Clinic, Vancouver, British Columbia
  - Clinique médicale Urbaine Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuel, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quigley A, Brouillette MJ, Fellows LK, Mayo N. Action for better brain health among people living with HIV: protocol for a randomized controlled trial. BMC Infect Dis. 2021 Aug 20;21(1):843. doi: 10.1186/s12879-021-06540-7. PMID 34416849